CLINICAL TRIAL: NCT02747667
Title: Late Dislocation and Haptic Deformation of a Hydrophilic Intraocular Lens: Characteristics, Incidence Rates and Predisposing Factors
Brief Title: Characteristics and Risk Ratios of Late Intraocular Lens (IOL) Complication
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Mayer Christoph, MD, MD, Medical University of Graz
Other Study IDs: 26-066 ex 13/14
Record Dates: First submitted 2016-04-17; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Complications
Keywords: iol dislocation; iol complication; intraocular lens; Implant or Graft; Eye

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eye with late IOL complication: Alle patients with IOL complication (subgroup: in-the-bag dislocation; out-of-the-bag dislocation; haptic dislocation)
- Eyes with no late IOl complication

SUMMARY:
Late in-the-bag intraocular lens (IOL) dislocation occurs up to 30 years after cataract surgery and the prevalence ranges from 0.1% to 3.0%. Before the introduction of the continuous curvilinear capsulorhexis, late dislocation was very uncommon but since then several case reports and case series were observed. In-the-bag IOL dislocation is a well-known postoperative complication, especially in eyes with weak zonules as seen in pseudoexfoliation syndrome (PXF), high axial myopia, uveitis and retinitis pigmentosa (RP).

In this retrospective study, medical records of all patients with IOL related problems after implantation of one hydrophilic acrylic single-piece lens at the Department of Ophthalmology Graz, Medical University Graz, Styria, Austria are reviewed. Characteristics and predisposing factors for late in-the-bag, out-of-the-bag IOL dislocations, and haptic complications will be investigated and compared amongst each other or control patients. Incidence rates for each IOL complication will be calculated. For in-the-bag dislocations odds ratios for each predisposing factor will be calculated.

DETAILED DESCRIPTION:
This is a retrospective cohort study. Data of all patients treated at the hospital from June 1997 to October 2015 for a complication after IOL implantation will be obtained from an electronic medical record and database (FileMaker Inc., v3 - 6 and EyMed). Additional data, e.g. axial length (AL) or diopters of the implanted IOL, are taken from the patients' medical files. Collected data are age, sex, laterality of the eye, and predisposing eye conditions (PXF, relevant myopia defined as ≥ 25.5 mm axial length, uveitis, RP and ocular trauma). Other parameters are preoperative surgical interventions, the use of a capsular tension ring (CTR), perioperative complications, diopters of the IOL, pre- and postoperative corrected distance visual acuity (CDVA) in logMAR, and post-operative manifest refraction. Time to dislocation, additional interventions after cataract surgery, and symptoms due to the IOL complication will recorded. Type of dislocation (in-the-bag or out-of-the-bag), location (anterior chamber, pupillary plane or vitreous), pre- and post-operative CDVA, pre- and post-operative manifest refraction, type of secondary intervention, and in case secondary implantation was performed, type of secondary IOL are collected.

Differences regarding prevalence for various predisposing risk factors are investigated by means of logistic regression methods. Odds ratios and 95% confidence intervals are calculated unadjusted as well as adjusted for age, gender, and the four predisposing risk factors: PXF, relevant myopia, uveitis, and RP. Prevalence and incidence of in-the-bag IOL dislocations will be calculated from all patients that had an implantation of the ACR6D SE at the Department of Ophthalmology in Graz.

ELIGIBILITY:
Inclusion Criteria:

* Phacoemulsification or extracapsular cataract extraction with the hydrophilic acrylic IOL ACR6D SE at the Department of Ophthalmology Graz in Styria, Austria.

Exclusion Criteria:

* Intracapsular cataract extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with phacoemulsification and extracapsular cataract surgery with the hydrophilic acrylic IOL ACR6D SE at the Department of Ophthalmology Graz in Styria, Austria.
Sampling Method: Non-Probability Sample
Enrollment: 10125 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of a late IOL complication (in-the-bag dislocation, out-of-the-bag dislocation and haptic bag dislocation) | 1997-2007 (retrospective)

SECONDARY OUTCOMES:
Incidence rates for a late IOL complication (in-the-bag dislocation, out-of-the-bag dislocation and haptic bag dislocation) | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor pseudoexfoliation (PXF) | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor myopia. | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor uveitis. | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor retinitis pigmentosa. | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor age. | 1997-2007 (retrospective)
Odds ratios for in-the-bag dislocations for predisposing risk factor sex. | 1997-2007 (retrospective)
Time from cataract operation to late in-the-bag dislocation. | 1997-2007 (retrospective)
Time from cataract operation to late out-of-the-bag dislocation. | 1997-2007 (retrospective)
Time from cataract operation to late haptic bending. | 1997-2007 (retrospective)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph F Mayer, MD, Principal Investigator — Medical University of Graz

IPD SHARING:
Plan to Share IPD: No